CLINICAL TRIAL: NCT03315169
Title: The Impact of Postoperative Packing of Perianal Abscess Cavities: a Multicentre Randomised Controlled Trial
Brief Title: Packing of Perianal Abscess Cavities
Acronym: PPAC2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: University of Liverpool (Other); Northwest Research Collaborative (Unknown); University of Birmingham (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R04689; PB-PG-0815-20037 (Other Grant/Funding Number: NIHR RfPB)
Record Dates: First submitted 2017-10-11; First posted 2017-10-20 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Perianal Abscess; Perianal Infections; Peri Rectal Abscess; Abscess; Anus; Abscess Anorectal
Keywords: Incision and Drainage; Packing
MeSH Terms: conditions — Abscess; Surgical Wound

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Note that only the clinician assessing healing and fistulae are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Packing of perianal abscess cavity (Active Comparator): Internal packing of perianal abscess cavity as per normal practice.
  Interventions: Other: Packing of perianal abscess cavity
- External dressing (Experimental): External application of a non-adherent dressing to the perianal abscess cavity.
  Interventions: Other: External dressing

INTERVENTIONS:
Other: External dressing — Application of external dressing whilst perianal abscess cavity heals.
  Arms: External dressing
Other: Packing of perianal abscess cavity — Internal packing of perianal abscess cavity - standard treatment.
  Arms: Packing of perianal abscess cavity

SUMMARY:
The aim of this trial is to compare internal wound packing to no packing in postoperative management following incision and drainage of perianal abscess. Participants will be randomised 1:1 to either the packing or non-packing arm.

DETAILED DESCRIPTION:
Perianal abscess is common, affecting 18,000 patients annually in England. Management has remained largely unchanged for over 50 years, and comprises surgical incision and drainage followed by continued internal wound dressing (packing) until healed. Packing is thought to reduce the rate of recurrent abscess and perianal fistula; a known complication of perianal abscess. Perianal fistula frequently requires multiple operations to resolve. The evidence for postoperative packing is limited¹ and may expose patients to painful procedures with no clinical benefit, and at considerable increased cost².

A multi-centre observational study of outcomes after drainage of perianal abscess (PPAC²) (n=141) found packing to be painful (2-3 fold increase in Visual Analogue Score pain scores during packing) and costly (estimated cost of £280 per patient; overall cost in the United Kingdom of £5 million annually). Fistula rate was 27%.

This study is a randomised controlled trial designed to assess whether there are differences between non-packing and packing of the perianal abscess cavity in terms of the short term negative effects of packing (pain, quality of life, return to work) whilst assessing the impact on key clinical outcomes (wound healing, fistulae formation) and resource use/cost.

All participants will be required to complete pain diaries following discharge from hospital. Clinical follow up to assess healing and other key clinical outcomes will take place at 4, 8 (if not healed at 4 weeks) and 26 weeks. Further data will be collected from National Health Service Registries at 52 weeks in order to assess abscess recurrences and fistulae formation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or over
2. Undergoing surgical incision and drainage of a primary perianal abscess

Exclusion Criteria:

1. Suspected inflammatory bowel disease
2. Fournier's Gangrene
3. Horseshoe (bilateral) abscess
4. Fistula-in-ano
5. Multiple abscess

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Wound-related pain intensity | Mean score over first 10 post-operative days
  Wound-related pain intensity (worst pain during previous 24 hours) measured using a single 100mm Visual Analogue Scale where 0 represents 'no pain' and 100 represents 'worst pain possible'. The pain Visual Analogue Scale is a continuous scale comprised of a horizontal line 100mm in length, anchored by 2 verbal descriptors, one for each symptom extreme, where 0 represents 'no pain' and 100 represents 'worst pain possible'. The mean score over the first 10 post-operative days will be used.

SECONDARY OUTCOMES:
Dressing-change related pain intensity | First 10 post-operative days
  Pain before, during and after dressing change measured using a 100mm Visual Analogue Scale where 0 represents 'no pain' and 100 represents 'worst pain possible'. The pain Visual Analogue Scale is a continuous scale comprised of a horizontal line 100 mm in length, anchored by 2 verbal descriptors, one for each symptom extreme. The mean score for each timepoint (before, during and after) over the first 10 post-operative days will be used.
Health related quality of life | On the 21st post-operative day
  Health related quality of life measured using EuroQol EQ-5D-5L quality of life questionnaires. The EQ-5D-5L descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension now has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The respondent is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions. This decision results in a 1-digit number expressing the level selected for that dimension. The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state.
Health utility | On the 21st post-operative day
  Health utility measured using EuroQol EQ-5D-5L quality of life questionnaires. The EQ-5D-5L descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension now has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The respondent is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions. This decision results in a 1-digit number expressing the level selected for that dimension. The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state.
Patient satisfaction with wound management | On the 21st post-operative day
  Patient satisfaction with wound management measured using a five point Likert scale. Patients are asked to mark the extent to which they agree with the statement 'I am satisfied with the way my wound has been treated following my surgery' where 1 equates to 'strongly disagree' and 5 equates to 'strongly agree'.
Rate of wound healing | Four and eight weeks post-operatively
  Rate of wound healing (complete epithelialization)
Clinical diagnosis of perianal abscesses recurrence after healing | 52 weeks post-operatively
  Clinical diagnosis of perianal abscesses recurrence after healing, ascertained either through clinical follow-up as part of trial procedures or via central National Health Service registries.
Chronic post-surgical pain | 4, 8 and 26 weeks post-operatively
  Chronic post-surgical pain measured using the Brief Pain Inventory - Short Form. The Brief Pain Inventory - Short Form assesses the severity of pain and the impact on daily functions. Pain is assessed at its "worst," "least," "average," and "now" (current pain), measured on a scale of 1-10 where 1 represents "no pain" and 10 represents "pain as bad as you can imagine". The four items will be represented singly but a composite of the four pain items (a mean score) will be presented as supplemental information. Pain interference (impact of pain on seven daily activities) will be scored as the mean of the seven interference items. These items are scored between 1 and 10, where 1 represents "does not interfere" and 10 represents "completely interferes".
Dressing use | Up to 52 weeks post-operatively
  Number of dressings used between time of operation up until week 52.
Health Professional contact time | Up to 52 weeks post-operatively
  Number of contacts with a Health Professional regarding perianal abscess or post-surgical complications between time of operation and 52 weeks post-operatively.
Hospital admission time | Up to 52 weeks post-operatively
  Number and length of hospital admissions as recorded in NHS central registries - Hospital Episodes Statistics.
Time to return to work or normal function | Up to 52 weeks post-operatively
  Length of time, measured in days, between operation and return to work or normal function.
Cost | Up to 52 weeks post-operatively
  Cost as applied to resource use data (see outcome 9-12)
Assessment of pain control methods | 21 days post-operatively
  Assessment of pain control methods (i.e. pain control medications) using Patient Global Assessment of the method of pain control where a rating of the pain control method over the past 24 hours is rated as being one of "poor," "fair," "good," or "excellent".
Fistula rate | Up ro 52 weeks post-operatively
  Fistula rate observed during clinical follow up and through Hospital Episodes Statistics

CONTACTS AND LOCATIONS:
Overall Officials: James Hill, FRCS, Principal Investigator — Manchester University NHS Foundation Trust
Locations (50):
- United Kingdom (50):
  - Salford Royal Hospital, Salford, Greater Manchester
  - West Middlesex University Hospital (Isleworth), Isleworth, Middlesex
  - John Radcliffe Hospital, Oxford, Oxfordshire
  - Mew Cross Hospital, Wolverhampton, West Midlands
  - Huddersfield Royal Infirmary, Huddersfield, West Yorkshire
  - Pindersfields General Hospital, Wakefield, West Yorkshire
  - Salisbury District Hospital, Salisbury, Wiltshire
  - Aberdeen Royal Infirmary, Aberdeen
  - Bangor Hospital, Betsi Cadwaladr University Health Board, Bangor
  - Furness General Hospital, Barrow in Furness
  - Royal United Hospital Bath NHS Foundation Trust, Bath
  - Birmingham Heartlands Hospital, Birmingham
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Royal Blackburn Hospital, Blackburn
  - Blackpool Victoria Hospital, Blackpool
  - Royal Bolton Hospital, Bolton
  - Bristol royal Infirmary, University Hospitals Bristol, Bristol
  - Southmead Hospital North Bristo; NHS Trust, Bristol
  - Addenbrooke's Hospital, Cambridge
  - University Hospital of Wales (Cardiff), Cardiff
  - Broomfield Hospital, Chelmsford
  - Countess of Chester, Chester
  - Chesterfield Royal Hospital NHS Foundation Trust, Chesterfield
  - University Hospitals Coventry and Warwickshire, Coventry
  - Royal Devon & Exeter Hospital, Exeter
  - Victoria Hospital (Fife), Kirkcaldy
  - Royal Lancaster Infirmary, Lancaster
  - Aintree Hospital, Liverpool
  - Royal Liverpool and Broadgreen University Hospitals NHS Trust, Liverpool
  - Royal Glamorgan Hospital, Llantrisant
  - Macclesfield District General Hospital, Macclesfield
  - Manchester Royal Infirmary, Manchester
  - Wythenshawe Hospital, Manchester
  - Queen Elizabeth The Queen Mother Hospital, Margate
  - Newcastle Upon Tyne University Hospitals NHS Foundation Trust, Newcastle
  - Royal Gwent Hospital, Newport
  - Norfolk and Norwich University Hospital, Norwich
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Royal Alexandra Hospital, Paisley
  - Plymouth Hospitals NHS Trust Derriford Hospital, Plymouth
  - Portsmouth Hospitals NHS Trust, Portsmouth
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Southampton General Hospital, Southampton
  - Arrowe Park Hospital, Upton
  - Warrington Hospital, Warrington
  - Warwick Hospital, South Warwickshire NHS Foundation Trust, Warwick
  - Sandwell Hospital, SWBH NHS Trust, West Bromwich
  - Royal Albert and Edward Infirmary, Wigan
  - Wrexham Maelor Hospital, Betsi Cadwaladr University Health Board, Wrexham
  - Yeovil District Hospital, Yeovil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith SR, Newton K, Smith JA, Dumville JC, Iheozor-Ejiofor Z, Pearce LE, Barrow PJ, Hancock L, Hill J. Internal dressings for healing perianal abscess cavities. Cochrane Database Syst Rev. 2016 Aug 26;2016(8):CD011193. doi: 10.1002/14651858.CD011193.pub2. PMID 27562822
- [Background] Pearce L, Newton K, Smith SR, Barrow P, Smith J, Hancock L, Kirwan CC, Hill J; North West Research Collaborative. Multicentre observational study of outcomes after drainage of acute perianal abscess. Br J Surg. 2016 Jul;103(8):1063-8. doi: 10.1002/bjs.10154. Epub 2016 Apr 7. PMID 27061287
- [Derived] Newton K, Dumville J, Briggs M, Law J, Martin J, Pearce L, Kirwan C, Pinkney T, Needham A, Jackson R, Winn S, McCulloch H, Hill J; PPAC2 Collaborators. Postoperative Packing of Perianal Abscess Cavities (PPAC2): randomized clinical trial. Br J Surg. 2022 Sep 9;109(10):951-957. doi: 10.1093/bjs/znac225. PMID 35929816